CLINICAL TRIAL: NCT05937620
Title: Sentinel Node Detection With Technetium-99m Albumin Nanocolloid and Indocyanine Green (ICG) in Patients With Epithelial Ovarian Cancer in Early Stages: Pilot Study
Brief Title: Sentinel Node Detection With Technetium-99m Albumin Nanocolloid and ICG in Patients With Epithelial Ovarian Cancer
Acronym: Melisa-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-505667-37-00
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional arm (Experimental): All patients will receive an injection of ICG and an injection of 99mTc nanocolloid albumin
  Interventions: Diagnostic Test: 99mTC nanocolloid albumin injection; Diagnostic Test: ICG injection

INTERVENTIONS:
Diagnostic Test: 99mTC nanocolloid albumin injection — All patients will receive an injection of both tracers in order to detect the sentinel lymph node
Diagnostic Test: ICG injection — All patients will receive an injection of both tracers in order to detect the sentinel lymph node

SUMMARY:
Study to evaluate the diagnostic precision of ICG and 99mTc nanocolloid albumin in sentinel lymph node detection in early ovarian epithelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adnexal mass diagnosed with high suspicion of malignancy that will undergo intraoperative biopsy or patients with already diagnosed epithelial cancer in early stages in a previous surgery and confirmed by pathology with complete staging indicated.
* Absence of retroperitoneal ganglionary affectation and metastatic disease evaluated by preoperative imaging techniques.
* Signing of informed consent by the patient or relative in charge.
* Women with childbearing potential must compromise to use highly effective contraceptive methods (partner vasectomized, sexual abstinence) until the end of the study (last study visit).

Exclusion Criteria:

* Patients <18 years
* Pregnancy or breastfeeding
* Epithelial ovarian tumors stage FIGO III or IV.
* Impossibility to obtain a biopsy from the tumor.
* History of previous vascular surgery (cava vein, aorta, iliac blood vessels) or radiotherapy in pelvic or para-aortic area.
* Sentinel lymph node biopsy will not be performed if intraoperative histologic study shows a benign ovarian tumor, low malignancy potential tumor or expansive mucinous histology.
* Patient not able to undergo surgery.
* Hypersensitivity to active principle, to sodium iodide or iodine allergy.
* Patients with clinic hyperthyroidism, thyroid autonomous adenomas or focal and diffused autonomous alteration of thyroid gland

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic efficiency of both tracers in sentinel lymph node detection | Through study completion (an average of 36 months)
  Global detection rate of sentinel lymph node in patients having received both tracers.

SECONDARY OUTCOMES:
Evaluation of diagnostic precision for the detection of sentinel lymph node detection in epithelial ovarian cancer in early stages according to morphological characteristics | Through study completion (an average of 36 months)
  Diagnostic precision defined as global detection rate of sentinel lymph nodes and false negatives rate, stratified by morphologic characteristics.
Evaluation of diagnostic precision for the detection of sentinel lymph node detection in epithelial ovarian cancer in early stages according to pathology results. | Through study completion (an average of 36 months)
  Diagnostic precision defined as global detection rate of sentinel lymph nodes and false negatives rate, stratified by pathology results
Evaluation of diagnostic precision for the detection of sentinel lymph node detection in epithelial ovarian cancer in early stages according to International Federation of Gynecology and Obstetrics (FIGO) stage | Through study completion (an average of 36 months)
  Diagnostic precision defined as global detection rate of sentinel lymph nodes and false negatives rate, stratified by FIGO stage
Evaluation of diagnostic precision for the detection of sentinel lymph node detection in epithelial ovarian cancer in early stages according to biochemistry results. | Through study completion (an average of 36 months)
  Diagnostic precision defined as global detection rate of sentinel lymph nodes and false negatives rate, stratified by biochemistry results
Evaluation of diagnostic precision for the detection of sentinel lymph node detection in epithelial ovarian cancer in early stages according to surgical approach | Through study completion (an average of 36 months)
  Diagnostic precision defined as global detection rate of sentinel lymph nodes and false negatives rate, stratified by surgical approach
Evaluation of anatomical distribution of 99mTC draining | Through study completion (an average of 36 months)
  Detection rate of sentinel lymph node with 99mTC in the group of patients having received the tracer
Evaluation of the performance of intraoperative detector gamma probe in the display of ovarian lymphatic map according to morphological characteristics. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative detector gamma probe,stratified by morphologic characteristics.
Evaluation of the performance of intraoperative detector gamma probe in the display of ovarian lymphatic map according to pathology results. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative detector gamma probe,stratified by pathology results.
Evaluation of the performance of intraoperative detector gamma probe in the display of ovarian lymphatic map according to FIGO stage. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative detector gamma probe,stratified by FIGO stage.
Evaluation of the performance of intraoperative detector gamma probe in the display of ovarian lymphatic map according to biochemistry results. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative detector gamma probe,stratified by biochemistry results.
Evaluation of the performance of intraoperative detector gamma probe in the display of ovarian lymphatic map according to surgical approach. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative detector gamma probe,stratified by surgical approach.
Evaluation of the performance of intraoperative Near Infrared (NIR) camera in the display of ovarian lymphatic map according to morphological characteristics | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative NIR camera,stratified by morphological characteristics
Evaluation of the performance of intraoperative NIR camera in the display of ovarian lymphatic map according to pathology results. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative NIR camera,stratified by pathology results.
Evaluation of the performance of intraoperative NIR camera in the display of ovarian lymphatic map according to FIGO stage. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative NIR camera,stratified by FIGO stage.
Evaluation of the performance of intraoperative NIR camera in the display of ovarian lymphatic map according to biochemistry results. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative NIR camera,stratified by biochemistry results.
Evaluation of the performance of intraoperative NIR camera in the display of ovarian lymphatic map according to surgical approach. | Through study completion (an average of 36 months)
  Detection rate and false negative rate of intraoperative NIR camera,stratified by surgical approach.
Anatomical distribution of sentinel lymph node detected with ICG. | Through study completion (an average of 36 months)
  Anatomical location of sentinel lymph node according to ICG.
Anatomical distribution of sentinel lymph node detected with 99mTC albumin nanocolloid. | Through study completion (an average of 36 months)
  Anatomical location of sentinel lymph node according to 99mTC albumin nanocolloid.
Comparison of lymph node detection with both tracers. | Through study completion (an average of 36 months)
  Assessment of concordance of sentinel lymph node anatomical location detected with each tracer.
Evaluation of ultra-staging in micrometastases detection compared to conventional histology. | Through study completion (an average of 36 months)
  Pathology ultra-staging evaluation.
  The following classification will be considered according to the criteria of the American Joint Committee on Cancer (AJCC):
  * Macrometastases: tumor infiltration > 2 mm in maximum diameter.
  * Micrometastases: tumor infiltration between 0.2 and 2 mm in maximum diameter.
  * Isolated tumor cells or isolated cell group (CTA, GCA): clusters of cells smaller than 0.2 mm
Evaluation of the complications associated with each technique. | Through study completion (an average of 36 months)
  Chirurgic and post-operative complications, directly or indirectly associated to the use of the tracers.

CONTACTS AND LOCATIONS:
Overall Officials: Berta Diaz-Feijoo, Physician, Principal Investigator — Hospital Clinic of Barcelona; Aureli Torné, Physician, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Laura Burunat, Barcelona, Catalonia, Spain